CLINICAL TRIAL: NCT01773499
Title: Sonographic Features of Cellulitis and Failure of Therapy
Status: Terminated | Type: Observational
Why Stopped: Unable to enroll significant number of patients.
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Romolo Gaspari, Associate Professor of Emergency Medicine, University of Massachusetts, Worcester
Other Study IDs: UMASSEDUS3
Record Dates: First submitted 2013-01-17; First posted 2013-01-23 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Cellulitis
Keywords: cellulitis; ultrasound
MeSH Terms: conditions — Cellulitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with Cellulitis: Patients with uncomplicated cellulitis treated as outpatients

SUMMARY:
Skin and soft tissue infections represent a tremendous burden to the health care community with over 11.6 million ambulatory patients presenting annually in 2003 and 14.2 million in 2005. A Cochrane review of cellulitis found that there is limited data to support any specific antibiotic or even a specific length of antibiotic therapy, and that outpatient therapy for cellulitis is increasing. Soft tissue ultrasound has been shown to have utility in differentiating cellulitis from abscess but its role in patients with cellulitis is not well developed. Although speculative, the investigators hypothesize that sonographic features of cellulitis are associated with clinical improvement and successful therapy following antibiotics for patients with cellulitis.

DETAILED DESCRIPTION:
The primary objective is to determine if changes in the sonographic features of cellulitis are associated with failure of therapy. Patients with cellulitis treated in the ED with either intravenous or oral antibiotics will undergo imaging using a standardized ultrasound protocol. Patients will be screened and enrolled in the ED at the UMASS Memorial Medical Center. The study design is single center prospective observational trial involving adult patients with clinical signs of cellulitis requiring antibiotics but not admitted to the hospital. Patients will be imaged upon initial presentation to the ED. Patients discharged from the ED after the initial visit will return to the ED in 24 to 48 hours for a reassessment. Patients kept in the ED under observational status will undergo an identical reassessment. Clinical staff blinded to the ultrasound results will characterize patients as improving, no change or worsening based on progression of the erythema despite antibiotics or change in clinical status. Researchers blinded to the clinical data will review the ultrasound images to quantify the extent of the sonographic evidence of cellulitis compared to the extent of the erythema by physical exam findings.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older Symptoms of cellulitis (localized warmth, erythema, swelling or tenderness)

Exclusion Criteria:

Admitted for inpatient antibiotics Unable to consent Septic appearing crepitus on exam animal bite soft tissue abscess osteomylitis cellulitis requiring surgical debridement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Cellulitis
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2013-01; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Failure of therapy | 7 days
  Patients with change in antibiotics or hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Romolo J Gaspari, MD, PhD, Principal Investigator — UMass Memorial Health
Locations (1):
- UMASS Memorial Medical Center, Worcester, Massachusetts, United States